CLINICAL TRIAL: NCT01384019
Title: Distal Protection Device Did Not Improve Microvascular Obstruction Evaluated by Cardiac MR After Primary Percutaneous Intervention for ST-elevation Myocardial Infarction
Brief Title: Distal Protection Device in ST-elevation Myocardial Infarction (STEMI)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Seoul National University Bundang Hospital (Other)
Responsible Party: Principal Investigator, Dong-Ju Choi, director of cardiovascular center, Seoul National University Bundang Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SNUBH-001
Record Dates: First submitted 2011-06-27; First posted 2011-06-28 (Estimated); Results first posted 2013-03-18 (Estimated); Last update posted 2013-03-18 (Estimated); Status verified 2013-02

CONDITIONS: ST-segment Elevation Myocardial Infarction
Keywords: ST-elevation myocardial infarction; percutaneous coronary intervention; cardiac magnetic resonance imaging; microvascular occlusion; myocardial salvage
MeSH Terms: conditions — ST Elevation Myocardial Infarction

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- DP-TA (Experimental): distal protection and thrombus aspiration during primary percutaneous coronary intervention (PCI) for ST-elevation myocardial infarction (STEMI)
  Interventions: Device: distal protection and thrombus aspiration (The GuardWire Plus (Medtronic Inc.))
- c-PCI (Placebo Comparator): conventional PCI without DP-TA during primary percutaneous coronary intervention for ST-elevation myocardial infarction
  Interventions: Procedure: c-PCI

INTERVENTIONS:
Device: distal protection and thrombus aspiration (The GuardWire Plus (Medtronic Inc.)) — The GuardWire Plus (Medtronic Inc.): distal balloon occlusion and proximal thrombus aspiration
  Other Names: The GuardWire Plus (Medtronic Inc.)
  Arms: DP-TA
Procedure: c-PCI — conventional PCI without Guard wire
  Other Names: convenional PCI
  Arms: c-PCI

SUMMARY:
The investigators examined the mechanism underlying the lack of benefit from distal protection and thrombus aspiration (DP-TA) in 126 patients with ST-elevation Myocardial Infarction (STEMI) in a prospective, randomized trial.

DETAILED DESCRIPTION:
Patients with first-diagnosed STEMI were randomly assigned to distal protection and thrombus aspiration (DP-TA) pretreatment during percutaneous coronary intervention (PCI) or conventional PCI (c-PCI).

The primary endpoint was the remodeling index (RI), measured by cardiac magnetic resonance imaging (CMR) post-PCI and 6 months after PCI.

Secondary endpoints, determined by CMR within 3 to 5 days after PCI, included the infarct ratio (infarct size to entire left ventricular [LV] size ) by delayed-enhancement (DE), area at risk (AAR) ratio (AAR to LV size) by T2 high-signal intensity , microvascular occlusion index (MVO) ratio (MVO to LV size) by DE, and myocardial salvage index (MSI, [AAR-infarct size] x 100/AAR).

ELIGIBILITY:
Inclusion Criteria:

* 30 and less than 80 years presenting with STEMI
* more than 30 minutes but less than 12 hours after symptom onset
* with ≥ 2 mm of ST-segment elevation in 2 or more contiguous leads or with a presumably new left bundle-branch block
* for whom primary PCI was intended

Exclusion Criteria:

* included thrombolytic therapy before PCI;
* spontaneous restoration of coronary flow (> TIMI grade II or III);
* cardiogenic shock (Killip class IV);
* major surgery or active bleeding within 6 weeks;
* aspirin, thienopyridine, or heparin allergy;
* neutropenia (<1000 neutrophils/mm3), thrombocytopenia (<100000 platelets/mm3), hepatic dysfunction, or renal insufficiency (serum creatinine level >2.5 mg/dL [221 μmol/L]);
* noncardiac condition with expected survival less than 1 year;
* current participation in other investigations.

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2004-01; Primary Completion 2008-06 (Actual); Study Completion 2011-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dong-ju Choi, MD, Principal Investigator — Seoul National University Bundang Hospital
Locations (1):
- Seoul Natioinal University Bundang Hospital, Seongnam, South Korea

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between Jan 24, 2004, and June 16, 2008, 550 patients with STEMI were screened.
Pre-assignment Details: Among them, 126 patients were randomized to receive either PCI with distal protection (n=65) or PCI alone (n=61). Fifty five patients per each group received post-PCI CMR. Forty one patients underwent 6 month MRI in distal protection group and 43 patients, in conventional PCI group.
Period: Overall Study
Arm/Group | DP-TA | c-PCI
Started | 65 | 61
Completed | 55 | 55
Not Completed | 10 | 6
Not completed — Withdrawal by Subject | 3 | 0
Not completed — Death | 1 | 0
Not completed — MRI refusal | 6 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | DP-TA | c-PCI | Total
Number analyzed (Participants) | 65 | 61 | 126
Age Continuous [Mean (Standard Deviation); unit: years] | 58 (12) | 58 (11) | 58 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 13 | 26
  Male | 52 | 48 | 100
Region of Enrollment [Number; unit: participants]
  Korea, Republic of | 65 | 61 | 126

OUTCOME MEASURES:

1. Primary Outcome: Postinfarct Remodeling
Description: postinfarct remodeling as evidenced by decreased left ventricular (LV) dilatation measured by CMR 6 months post PCI
Time Frame: 6 months
Population: Forty one patients underwent 6 month CMR in distal protection group and 43 patients, in conventional PCI group.
Measure: Number; unit: Number of participants with remodeling
Arm/Group | DP-TA | c-PCI
Number analyzed (Participants) | 41 | 43
Number of participants with remodeling | 11 | 6

2. Secondary Outcome: Reperfusion Success
Description: microvascular obstruction, myocardial salvage, and infarct size measured using post-PCI CMR
Time Frame: 3-5 days
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | DP-TA | c-PCI
Serious Adverse Events (participants affected / at risk) | 7/65 | 7/61
Other Adverse Events (participants affected / at risk) | 0/65 | 0/61
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DP-TA (N=65) | c-PCI (N=61)
Death (Cardiac disorders) | 1 (1) | 2 (2)
revascularization (Cardiac disorders) | 6 (6) | 4 (4)
stroke (Cardiac disorders) | 0 (0) | 1 (1)
admission due to heart failure (Cardiac disorders) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No